CLINICAL TRIAL: NCT06366113
Title: Effect of Time of Exercise Re-training on Functional Capacity in Individuals With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Time of Exercise Re-training With Chronic Obstructive Pulmonary Disease (COPD)
Acronym: CHRONOBIO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michaël RACODON (Other)
Responsible Party: Sponsor-Investigator, Michaël RACODON, Head of clinical research, Clinique de la Mitterie
Organization: Clinique de la Mitterie (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-A00363-42
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Diseases
Keywords: respiratory diseases; pulmonary rehabilitation; chronic obstructive pulmonary disease; biological clock
MeSH Terms: conditions — Respiratory Tract Diseases; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning group (Other): Endurance and muscular exercise can be performed in the morning, either at 9:00am or 9:45am, or vice versa.
  Interventions: Other: Pulmonary rehabilitation
- Afternoon group (Other): Endurance and muscular exercise can be performed in the afternoon, from 3:00 pm to 3:45 pm, or vice versa.
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: Pulmonary rehabilitation — Pulmonary rehabilitation includes :
  * Exercise re-training with resumption of physical activities
  * therapeutic patient education

SUMMARY:
Pulmonary rehabilitation (PR) is an effective intervention for reducing hospital readmissions, secondary events, and mortality in patients with respiratory pathologies.

The program should not be improved by introducing new subjects such as circadian rhythm.

DETAILED DESCRIPTION:
Respiratory diseases are a leading cause of death in developed countries. To avoid complications and recurrences, secondary prevention in patients with respiratory diseases is essential. Pulmonary rehabilitation (PR) is a well-established and effective treatment that is supervised by medical professionals and conducted in dedicated centres. It has been shown to reduce hospital readmissions, secondary events, and patient mortality.

The timing of reconditioning is crucial. Previous studies have indicated that training times affect strength and power gains. Additionally, the time of day for training can significantly impact progress in aerobic capacity.

Disturbances to the biological clock can have consequences for people with respiratory pathologies, particularly an alteration in muscular function.

Therefore, studying the temporal specificity of exercise re-training in patients with respiratory diseases is of interest.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient with chronic obstructive pulmonary disease (COPD)
* Registered for respiratory re-education and rehabilitation at the Clinique de la Mitterie
* Number of rehabilitation sessions at least 18 over 4 weeks
* Written informed consent signed by the patient
* Membership of a social security

Exclusion Criteria:

* - cardiovascular contraindications to exercise
* unstable respiratory status (uncompensated respiratory acidosis)
* conditions interfering with the pulmonary rehabilitation process (progressive neuromuscular disease, psychiatric illness)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
6-minute walk test (6MWT) | 15 minutes
  Walking distance in a test

SECONDARY OUTCOMES:
Time limit test (Time-lim) | 0 to 900 secondes
  Endurance exercise holding time in seconds
Sit to stand test (STT) | 1 minute
  The number of sit-to-stand repetitions during the test.
Single arm curl Test (SAC) | 1 minute
  The number of bends during the test
Single-leg stance test (SLT) | 1 minute
  The time for balance
Hospital Anxiety and Depression Scale (HAD) | 10 minutes. The maximum mark for each score is 21 and the minimum mark is 0. The higher the score, the more depressed or anxious the person.
  Hospital Anxiety and Depression score
Pittsburgh Sleep Quality Index | 10 minutes. The total score ranges from 0 to 21, with 0 indicating no difficulties and 21 indicating major difficulties.
  Sleep quality score

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique la Mitterie, Lille, France

IPD SHARING:
Plan to Share IPD: Undecided
The IPD sharing plan with other researchers is only available on site at the clinic.